CLINICAL TRIAL: NCT03822091
Title: Comparison of The Effectiveness of Terlipressin Infusion Alone Vs Terlipressin With Noradrenaline Infusion In The Treatment of Hepatorenal Syndrome Type 1
Brief Title: Terlipressin Infusion Alone Vs Terlipressin With Noradrenaline Infusion In The Treatment of Hepatorenal Syndrome Type 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TERLI AND NORAD IN HRS
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Type 1 HEPATO RENAL SYNDROME(HRS)
MeSH Terms: interventions — Terlipressin; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TERLIPRESSIN GROUP (Active Comparator)
  Interventions: Drug: Terlipressin
- TERLIPRESSIN WITH NORADRENALINE GROUP (Experimental)
  Interventions: Drug: Terlipressin and Noradrenaline

INTERVENTIONS:
Drug: Terlipressin — Patients with Type 1 HRS will be given Terlipressin at the dose of 2mg/24 hrs as infusion. After 48 hours of initial monitoring, patients who do not respond to the initial dose of Terlipressin, and randomised into group A and B. Group A patients will receive further higher doses of Terlipressin. The dose of Terlipressin will be increased by 1mg after 24 hrs if:
  * the creatinine values decrease by <12.5%
  * MAP increase of <10 mmHg
  * urine output of <200 ml in 4 hours.
  Maximum terlipressin dose will be given upto 12 mg/day.Albumin will be administered in both arms according to standard protocol at the following dose :
  1. 1st day - Albumin at 1 gram/kg - a maximum dose of 100grams can be given.
  2. A dose of 20gram/day to 60gram/day in the following days.
  Arms: TERLIPRESSIN GROUP
Drug: Terlipressin and Noradrenaline — Patients with Type 1 HRS will be given Terlipressin at the dose of 2mg/24 hrs as infusion. After 48 hours of initial monitoring, patients who do not respond to the initial dose of Terlipressin, will be randomised into group A and B. Group B patients will be treated with
  Terlipressin(2mg/24hr infusion- fixed dose) and Noradrenaline, which would be given as a continuous infusion at a starting dose of 0.5 mg/hr. The dose od noradrenaline will be increased every 24 hours in steps of 0.5 mg/hr, the maximum dose being 3 mg/hr IF:
  * the creatinine values decrease by <12.5%
  * MAP increase of <10 mmHg
  * urine output of <200 ml in 4 hours.
  Arms: TERLIPRESSIN WITH NORADRENALINE GROUP

SUMMARY:
Hepatorenal syndrome (HRS) is defined as a functional renal failure in a patient with chronic liver disease, or liver cirrhosis.The splanchnic circulation undergoes severe vasodilation, as a result of portal hypertension, causing an underfilling of systemic arteries.This results in intense renal vasoconstriction and functional renal failure. The best treatment options for HRS I would be a drug which has renal vasodilator property and additional splanchnic vasoconstriction. An increase in circulating blood volume would be of additional benefit. Currently Terlipressin is considered superior to other drugs in the management of HRS I. Other drugs in use are Noradrenaline and Midodrine. Albumin is added to these drugs in order to expand plasma volume. Terlipressin, a Vasopressin analog, has agonistic activity at V1 receptors. Noradrenaline acts as an agonist at α-adrenergic receptors with mild β-agonistic activity. The two major drugs used in the management of HRS act at different receptors and have completely varied mechanisms of action. Thus, a combination therapy would improve the rate of response considerably. There have been multiple studies, measuring the efficacy, safety and dosing of both drugs, but none combining both Terlipressin and Noradrenaline. Hence our study would be a pioneer in formulating a new and possibly more efficacious treatment protocol for patients of Type I HRS, in whom the treatment options are otherwise very limited. If successful, this would open new horizons of therapy for Terlipressin refractory HRS, which, otherwise is an ominous condition.

ELIGIBILITY:
Inclusion Criteria:

1. age>18 years and <80 yrs;
2. Cirrhosis as diagnosed by clinical findings, endoscopy or USG examination or by liver biopsy.
3. HRS I as defined by the following features:

   1. The patient should have Cirrhosis and also ascites
   2. Renal failure of rapid onset -Initial value of sCr, doubling to reach a level of more than 226mmol/L (2.5 mg/dL) in less than two weeks
   3. There should be absence of shock.
   4. sCr value does not reduce to less than 1.5 mg/dl even after 2 days of stopping diuretics and giving Inj.Albumin for plasma volume expansion (1g/kg ) upto 100g/day.
   5. No H/O being treated currently or recently with drugs having nephrotoxicity.
   6. Absence of parenchymal renal disease:

      * Proteinuria < 0.5g/day
      * Absence of microhaematuria (<50 red cells/high powered field)
      * Normal renal ultrasonography

Exclusion Criteria:

1. AKI improved after plasma volume expansion
2. Any history of coronary artery disease, peripheral vascular disease, arrhythmias, and cardiomyopathy.
3. Hepatocellular Carcinoma
4. Septic shock
5. Any severe extra-hepatic condition including respiratory and cardiac failure.
6. Any contraindication which precludes the use of Noradrenaline and Terlipressin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Number of patients responding to treatment. | 15 days
  Complete response defined as serum creatinine <1.5 mg/dl

SECONDARY OUTCOMES:
Number of patients who will develop adverse events due to drugs used for treatment | 15 days
Number of patients surviving without transplant. | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh V, Jayachandran A, De A, Singh A, Chandel S, Sharma N. Combination of terlipressin and noradrenaline versus terlipressin in hepatorenal syndrome with early non-response to terlipressin infusion: A randomized trial. Indian J Gastroenterol. 2023 Jun;42(3):388-395. doi: 10.1007/s12664-023-01356-6. Epub 2023 May 5. PMID 37145232